CLINICAL TRIAL: NCT05026320
Title: Randomized, Controlled, Double-blind, Placebo-controlled, Multi-center Hypothesis-finding Trial to Compare the Efficacy and Safety of a 10% Naproxen Gel vs. a 2.32% Diclofenac Diethylamine Gel and Placebo in the Treatment of Acute Soft Tissue Injuries of the Lower Extremities
Brief Title: A Clinical Trial to Compare Safety and Effectiveness for Relieving Tenderness of 10% Naproxen Gel vs. a 2.32% Diclofenac Diethylamine Gel in the Treatment of Strains and Bruises of the Legs.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Deutsche Sporthochschule Köln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21559; 2020-004343-92 (EudraCT Number)
Record Dates: First submitted 2021-07-12; First posted 2021-08-30 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Soft Tissue Injury
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Naproxen Topical Gel (BAYH006689) (Experimental): UI Number: 1614000-268; Subjects will be randomized into one of the three treatment groups in a 2:2:1 (active:active:placebo) allocation. Treatment consists of a twice daily (bid) application (approximately 12 hours apart) of the assigned topical gel over 5 consecutive days, beginning on the evening of Day 1 and ending (last application) on the morning of Day 6 (total of 10 applications). In order to assure adequate representation of different types of soft tissue injuries, at least 25 randomized subjects must enter the study with a lower extremity sprain/strain injury (cohort) and at least 50 randomized subjects with a lower extremity contusion injury (cohort).
  Interventions: Drug: Naproxen gel
- Diclofenac Diethylamine Gel (Active Comparator): UI Number: Not applicable; Subjects will be randomized into one of the three treatment groups in a 2:2:1 (active:active:placebo) allocation. Treatment consists of a twice daily (bid) application (approximately 12 hours apart) of the assigned topical gel over 5 consecutive days, beginning on the evening of Day 1 and ending (last application) on the morning of Day 6 (total of 10 applications). In order to assure adequate representation of different types of soft tissue injuries, at least 25 randomized subjects must enter the study with a lower extremity sprain/strain injury (cohort) and at least 50 randomized subjects with a lower extremity contusion injury (cohort).
  Interventions: Drug: Diclofenac gel
- Placebo Gel (Placebo Comparator): UI Number: 1614000-272; Subjects will be randomized into one of the three treatment groups in a 2:2:1 (active:active:placebo) allocation. Treatment consists of a twice daily (bid) application (approximately 12 hours apart) of the assigned topical gel over 5 consecutive days, beginning on the evening of Day 1 and ending (last application) on the morning of Day 6 (total of 10 applications). In order to assure adequate representation of different types of soft tissue injuries, at least 25 randomized subjects must enter the study with a lower extremity sprain/strain injury (cohort) and at least 50 randomized subjects with a lower extremity contusion injury (cohort).
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Naproxen gel — 10%, bid for 5 days (final application on morning of Day 6)
  Arms: Naproxen Topical Gel (BAYH006689)
Drug: Diclofenac gel — 2.32% bid for 5 days (final application on morning of Day 6)
  Arms: Diclofenac Diethylamine Gel
Drug: Placebo gel — bid for 5 days (final application on morning of Day 6)
  Arms: Placebo Gel

SUMMARY:
Researchers are looking for a different way to treat people who have an injury to their muscles, ligaments, or tendons in their legs or feet. This is known as a "soft tissue" injury. Before a treatment is available to all patients, researchers study it in trials to better understand its safety and how well it works.

People with soft tissue injuries can have pain, swelling, and bruising.

In this trial, the researchers want to learn more about the trial treatment, BAYH006689, in participants with a soft tissue injury to their legs or feet. BAYH006689 is a naproxen gel that is used for the temporary relief of minor aches and pains of muscles and joints. The researchers will learn more about how BAYH006689 works and how safe it is in these participants.

The trial will include about 100 male and female participants between the ages of 18 and 60. All the participants will have a soft tissue injury to their legs or feet that was caused by playing sports. The injury will have happened within 3 hours of joining the trial.

The researchers will use a computer program to randomly choose what treatment each participant will receive. This will help make sure the treatments are chosen fairly and that comparing the results of the treatments is as accurate as possible. The participants will be randomly chosen to be in 1 of 3 groups:

* Group 1: BAYH006689
* Group 2: diclofenac diethylamine gel
* Group 3: placebo

A placebo looks like a treatment but does not have any medicine in it. Diclofenac diethylamine gel is a treatment already available for doctors to be recommended to people with soft tissue injuries. The participants will receive their treatment once in the evening on Day 1 and then 2 times a day for 4 days. The participants will receive their final dose in the morning of Day 6. The doctors will apply the treatment to the participants' skin where the injury is.

The participants must be present at the clinic site 11 times over six days: once on Day 1 and twice daily on Days 2-6. During the trial, the doctors will:

* check the participants' overall health and ask if they have any medical problems
* do physical examinations to check the participants' injuries
* use a device to see how tender and sore the participants' injuries are

In this trial, the researchers will study how tender the participants' injuries are after 3 days and at other time points over the 6 day follow-up period. They will also study how many participants have medical problems during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 60 years of age inclusive, at the time of signing the informed consent.
* Participants with a primary diagnosis of acute sports-related acute soft tissue injuries of the lower extremities that do not require hospitalization and that occurred within 3 hours of enrollment.
* Participants with a baseline algometric measurement values on the injured site of ≤50% of the respective value at the contralateral site.
* Participants with a baseline pain on movement (POM) of ≥50 mm on a visual analog scale (VAS) (0-100 mm).
* Participant's absolute sensitivity to tenderness on the contralateral site is at least 2.5 N/cm2 as measured by algometry.
* Participant's size of trauma is between 25 and 150 cm^2.

Exclusion Criteria:

* Heart surgery within 2 weeks of enrollment in the study.
* Suspected bone fracture or torn ligaments related to the injury.
* Open wounds to the area to be treated.
* Current skin disorders or localized infection in the area to be treated.
* Injured area is too hairy for proper assessments.
* Suspected head injury.
* History of blood coagulation disorders.
* Current or past history of gastrointestinal ulceration, gastrointestinal bleeding or other bleeding disorder(s).
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted).
* History of significant disease deemed by the investigator to render the patient unsuitable for inclusion, including evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension and cardiac arrhythmia), hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years.
* Participants with a medical disorder, condition, or history of such that could impair the participant's ability to participate or complete this trial in the opinion of the investigator.
* Significant ongoing painful condition other than that associated with the sports-related injury/contusion.
* Any ongoing condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication.
* Females who are planning to become pregnant, are pregnant or lactating. Prior/Concomitant Therapy
* Ice and compression are prohibited from the time of injury through the final evaluation.
* Physical therapy or other comfort measures, or herbal preparations for bruises from the time of injury through the final evaluation.
* Use of any medications within 5 days of enrollment until discharge from the study site (except oral contraceptives, prophylactic antibiotics, synthetic thyroid hormones, methylphenidate or medications to treat benign conditions such as antibiotics to treat acne).
* Any other treatment or medication (oral or topical), that could interfere with the trial (e.g. corticosteroids) up to 3 days prior to the trial.
* Participants with the following medical conditions may be eligible at the discretion of the investigator: ADHD on a stable dose regimen of methylphenidate/(dextro) amphetamine for at least 6 months; participants with hypothyroidism on a stable dose of synthetic thyroid hormone for at least 6 months.
* Have received any form of treatment in the form of medication for depression in the past 6 months or any form of psychotropic agent (including selective serotonin uptake inhibitors [SSRI] but excluding ADHD medications described above) within the last 6 months.
* Any previous history of allergy or known intolerance to naproxen, diclofenac, paracetamol or any of the drugs or formulation constituents which, in the investigator's opinion, might preclude use of an NSAID, including aspirin-sensitive asthma or a previous allergic response to a NSAID, including bronchospasm, urticaria, angioedema, and rhinitis; participation in a clinical trial in the previous 30 days.
* Use of any over the counter (OTC) or prescription medications with which the administration of naproxen, acetaminophen, any other NSAID, is contraindicated.
* Habituation to analgesic drugs including opioids (i.e., routine use of oral analgesics 5 or more times per week for greater than 3 weeks within the past 2 years).

Other Exclusions

* More than low-risk alcohol consumption (>24 g (males) or ˃12 g (females) of alcohol regularly per day). Amount corresponds to 0.6 L of beer/day or 0.24 L of wine/day or 3 glasses (at 2 cL) of liquor/day for males and 0.3 L of beer/day or 0.12 L of wine/day or 1 glass (at 2 cL) of liquor/day for females.
* Self-reported drug abuse within two years prior to screening.
* Member or first-degree relative of study staff or the Sponsor directly involved in the study.
* Unwilling or unable to comply with all requirements outlined in the protocol.
* Previous enrollment in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsche Sporthochschule Köln (DSHS), Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in three centers in Germany. First participant first visit of the study was on 08 AUG 2021, and last participant last visit was on 20 DEC 2021.
Pre-assignment Details: Overall 76 participants completed screening and were randomized.
Groups:
- Naproxen Topical Gel: Participants received naproxen topical gel twice daily for 5 days.
- Diclofenac Diethylamine Topical Gel: Participants received diclofenac diethylamine topical gel twice daily for 5 days.
- Placebo: Participants received placebo twice daily for 5 days.
Period: Overall Study
Arm/Group | Naproxen Topical Gel | Diclofenac Diethylamine Topical Gel | Placebo
Started (76) | 31 | 30 | 15
Completed (76) | 31 | 30 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Topical Gel | Diclofenac Diethylamine Topical Gel | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 15 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.32 (10.74) | 31.57 (9.47) | 32.47 (13.05) | 32.46 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 9 | 41
  Male | 15 | 14 | 6 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 29 | 30 | 15 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic/Latino | 21 | 19 | 10 | 50
  Other | 9 | 11 | 5 | 25
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tenderness (Algometry) Over the Initial 72 Hours
Description: Algometry area under the curve (AUC) from zero to the initial 72h post dose. The 72h AUC algometry data was an aggregate of all measurements from timepoints and data including the 72h timepoint. The average data of all participants was reported.
Time Frame: Up to the initial 72 hours post dose
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Nxh/cm^2
Arm/Group | Naproxen Topical Gel | Diclofenac Diethylamine Topical Gel | Placebo
Number analyzed (Participants) | 30 | 28 | 14
Nxh/cm^2 | 1213.88 (461.11) | 1041.04 (274.25) | 850.79 (276.04)
Statistical Analysis 1: Comparison: Naproxen Topical Gel vs Diclofenac Diethylamine Topical Gel vs Placebo; Test type: Equivalence — The primary efficacy hypothesis to be tested was the equality of tenderness (algometry) over the initial 72 hours (algometry AUC 0-72); p = 0.0221, ANCOVA

2. Secondary Outcome: Percentage of Participants With at Least One Treatment Emergent Adverse Event After Treatment
Description: An AE is any untoward medical occurrence in a clinical study participant, associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: After first treatment on Day 1 until follow-up visit (Day 30)
Population: Safety population
Measure: Number; unit: Percentage
Arm/Group | Naproxen Topical Gel | Diclofenac Diethylamine Topical Gel | Placebo
Number analyzed (Participants) | 31 | 30 | 15
Percentage
  any AE | 0 | 3.33 | 0
  serious AE | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event After Treatment
Description: as for outcome 2
Time Frame: After first treatment on Day 1 until follow-up visit (Day 30)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Topical Gel | Diclofenac Diethylamine Topical Gel | Placebo
Number analyzed (Participants) | 31 | 30 | 15
Participants
  Rhinitis | 0 | 1 | 0
  Nasal congestion | 0 | 1 | 0
  Paranasal sinus hypersecretion | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after first treatment on Day 1 until follow-up visit (Day 30).
Groups:
- Naproxen Gel: Participants received Naproxen topical gel (BAYH006689) two times a day (bid) for 5 days.
- Diclofenac Gel: Participants received Diclofenac Diethylamine gel bid for 5 days.
- Placebo Gel: Participants received Placebo gel bid for 5 days.
Arm/Group | Naproxen Gel | Diclofenac Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 0/31 | 1/30 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Gel (N=31) | Diclofenac Gel (N=30) | Placebo Gel (N=15)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecret (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) agrees to submit any proposed publication, abstract or presentation related to the Study ("Publication") to Sponsor at least 30 days prior to submission. Sponsor shall advise PI or Designee in writing of any information that is Confidential Information (CI) or Sponsor's Intellectual Property (SIP). Sponsor shall have the right to require PI or Designee, to remove CI and/or delay the Publication for an additional 60 days to enable Sponsor to seek protection of SIP.

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT05026320/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT05026320/SAP_001.pdf